CLINICAL TRIAL: NCT00964431
Title: A Phase 2, Randomized, Double-Blind, Single-Dose, Parallel-Group, Active- and Placebo-Controlled Study of Indomethacin Test Capsules for the Treatment of Pain After Surgical Removal of Impacted Third Molars
Brief Title: Phase 2 Study of Indomethacin Capsules to Treat Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IND2-08-03
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-03

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Indomethacin Test (lower dose) (Experimental)
  Interventions: Drug: Indomethacin Test (lower dose)
- Indomethacin Test (upper dose) (Experimental): Single dose
  Interventions: Drug: Indomethacin Test (upper dose)
- Celecoxib 400 mg (Active Comparator)
  Interventions: Drug: Celecoxib 400 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib 400 mg — Capsules 2 x 200 mg Single-Dose
  Arms: Celecoxib 400 mg
Drug: Placebo — Capsules 2 Single-Dose
  Arms: Placebo
Drug: Indomethacin Test (lower dose) — 20-mg single dose
  Arms: Indomethacin Test (lower dose)
Drug: Indomethacin Test (upper dose) — 40-mg single dose
  Arms: Indomethacin Test (upper dose)

SUMMARY:
The purpose of this study is to determine whether Indomethacin Test Formulation Capsules are safe and effective for the treatment of dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 50 years of age
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Patient requires extraction of 2 or more third molars
* Patient must be willing to stay at the study site for at least 8 hours after dosing of the study drug

Exclusion Criteria:

* Patient has hypersensitivity, allergy, or clinically significant intolerance to any medications to be used in the study, or related drugs
* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen or alcohol breathalyzer test
* Patient has taken another investigational drug within 30 days prior to Screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Premier Research Group Limited, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indomethacin Test (Lower Dose) | Indomethacin Test (Upper Dose) | Celecoxib 400 mg | Placebo
Started | 50 | 51 | 51 | 51
Completed | 50 | 51 | 51 | 51
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indomethacin Test (Lower Dose) | Indomethacin Test (Upper Dose) | Celecoxib 400 mg | Placebo | Total
Number analyzed (Participants) | 50 | 51 | 51 | 51 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 51 | 51 | 51 | 203
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.0 (3.32) | 22.2 (3.81) | 22.1 (3.46) | 22.1 (2.97) | 22.1 (3.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 34 | 35 | 132
  Male | 18 | 20 | 17 | 16 | 71
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 51 | 51 | 203

OUTCOME MEASURES:

1. Primary Outcome: Total Patient Pain Relief Over 0 to 8 Hours.
Description: Total patient pain relief was assessed as a time-weighted sum of the patient pain assessments at each individual time point from 0-8 hours.
  Values for TOTPAR are measured from 0 to 4 on the Pain Relief Scale 0 None Min; 1 A little; 2 Some; 3 A lot; 4 Complete Max
  The TOTPAR is a weighted measure of the observations; the minimum possible value is 0 and the maximum possible value is 32.
Time Frame: 8 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Indomethacin Test (Lower Dose): 20-mg
- Indomethacin Test (Upper Dose): 40-mg
Arm/Group | Indomethacin Test (Lower Dose) | Indomethacin Test (Upper Dose) | Celecoxib 400 mg | Placebo
Number analyzed (Participants) | 50 | 51 | 51 | 51
units on a scale | 10.794 [8.131 to 13.456] | 12.564 [9.928 to 15.200] | 14.822 [12.185 to 17.460] | 3.019 [0.381 to 5.656]
Statistical Analysis 1: Comparison: Indomethacin Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 9.545, 95% CI 2-sided [5.816 to 13.275], Standard Error of Mean 1.8912

ADVERSE EVENTS:
Arm/Group | Indomethacin Test (Lower Dose) | Indomethacin Test (Upper Dose) | Celecoxib 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 19/50 | 26/51 | 19/51 | 29/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indomethacin Test (Lower Dose) (N=50) | Indomethacin Test (Upper Dose) (N=51) | Celecoxib 400 mg (N=51) | Placebo (N=51)
Alveolar osteitis (Gastrointestinal disorders) | 2 | 5 | 5 | 4
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 4
Headache (Nervous system disorders) | 3 | 4 | 4 | 8
Nausea (Nervous system disorders) | 8 | 6 | 5 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 3 | 5 | 3 | 4
Vomiting (Gastrointestinal disorders) | 2 | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No